CLINICAL TRIAL: NCT03368664
Title: A Multi-center, Open-label, Single-arm, Before and After Switch Study to Evaluate the Efficacy, Safety and Tolerability of Alemtuzumab in Paediatric Patients With Relapsing Remitting Multiple Sclerosis (RRMS) With Disease Activity on Prior Disease Modifying Therapy (DMT)
Brief Title: A Study to Evaluate Efficacy, Safety, and Tolerability of Alemtuzumab in Pediatric Patients With RRMS With Disease Activity on Prior DMT
Acronym: LemKids
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrolment formally closed earlier than planned due to recruitment challenges.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC13429; U1111-1180-6352 (Registry Identifier: ICTRP); 2016-003100-30 (EudraCT Number)
Record Dates: First submitted 2017-11-02; First posted 2017-12-11 (Actual); Results first posted 2022-07-12 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Alemtuzumab; Glatiramer Acetate; Interferon-beta; Methylprednisolone; Ranitidine; ceterizine hydrochloride; dexchlorpheniramine; Acetaminophen; Acyclovir; Prednisolone; aminophylline, cycloclenbutrerol, diphenydramine, phenobarbital drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Alemtuzumab (Experimental): - alemtuzumab - Dose 1 (initial course) of alemtuzumab will be administered intravenously on 5 consecutive days, followed by Dose 2 (second course) on 3 consecutive days administered 12 months after initial course. Pre-medications (methylprednisolone, prednisolone, H1 antagonist [antihistamine], H2 antagonist, paracetamol, acyclovir) will be administered prior alemtuzumab administration. - Type: Experimental
  Interventions: Drug: Alemtuzumab GZ402673; Drug: Glatiramer acetate; Drug: Beta-Interferon; Drug: Methylprednisolone; Drug: Ranitidine; Drug: Ceterizine; Drug: Dexchlorpheniramine; Drug: Paracetamol; Drug: Acyclovir; Drug: Prednisolone; Drug: Diphenydramine; Drug: Other H1 antagonist

INTERVENTIONS:
Drug: Alemtuzumab GZ402673 — Pharmaceutical form: solution, Route of administration: IV
  Other Names: Lemtrada
Drug: Glatiramer acetate — Pharmaceutical form: solution, Route of administration: subcutaneous (SC)
  Other Names: Copaxone
Drug: Beta-Interferon — Pharmaceutical form: solution, Route of administration: SC / intramuscular (IM)
Drug: Methylprednisolone — Pharmaceutical form: solution, Route of administration: IV
Drug: Ranitidine — Pharmaceutical form: tablet, Route of administration: oral
Drug: Ceterizine — Pharmaceutical form: tablet, Route of administration: oral
Drug: Dexchlorpheniramine — Pharmaceutical form: tablet, Route of administration: oral
Drug: Paracetamol — Pharmaceutical form: tablet, Route of administration: oral
Drug: Acyclovir — Pharmaceutical form: tablet, Route of administration: oral
Drug: Prednisolone — Pharmaceutical form: tablet, Route of administration: oral
Drug: Diphenydramine — Pharmaceutical form: solution, Route of administration: IV
Drug: Other H1 antagonist — Pharmaceutical form: solution, Route of administration: IV
Drug: Other H1 antagonist — Pharmaceutical form: tablet/pill, Route of administration: oral

SUMMARY:
Primary Objective:

To evaluate the efficacy, safety, and tolerability of alemtuzumab intravenously (IV) in pediatric participants from 10 to less than (<) 18 years of age with Relapsing Remitting Multiple Sclerosis (RRMS) who have disease activity on prior DMT.

Secondary Objective:

To assess the pharmacokinetics (PK), pharmacodynamics (PD), anti-drug antibody (ADA) formation, and potential effects of alemtuzumab on other multiple sclerosis (MS) disease characteristics such as cognition and quality of life (QoL).

DETAILED DESCRIPTION:
The duration of study per participant will be approximately 5 years and 5 months.

ELIGIBILITY:
Inclusion criteria :

* Participants with RRMS aged from 10 years to <18 years at study entry are eligible. Participants must meet the criteria of diagnosis of MS as defined by the International Pediatric MS Study Group (IPMSSG) criteria for pediatric MS and the criteria of MS based on 2010 McDonald criteria.
* Signed written informed consent/assent obtained from participant and participant's legal representative (parent or guardian) according to local regulations.
* Expanded Disability Status Scale (EDSS) score of 0.0 to 5.0 (inclusive) at screening.
* At least 2 recorded MS attacks and at least 1 MS attack (relapse) in the last year during treatment with a beta interferon therapy (IFNB) or glatiramer acetate (GA) after being on that therapy for at least 6 months, and was currently still taking the same therapy.
* At least 1 of the following:
* >=1 new or enlarging T2 hyperintense lesion or gadolinium enhancing lesion while on that same prior therapy (IFNB or GA), or
* Two or more relapses in the prior year, or
* Tried at least 2 MS DMTs.

Exclusion criteria:

* Any progressive or non-relapsing forms of MS.
* Conditions/situations such as:
* Impossibility to meet specific protocol requirements.
* Current participation in another interventional clinical study. Participants who are treated with a comparator agent approved for screening inclusion (INF or GA) may be considered for this trial.
* Participant is the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
* Uncooperative participant or any condition that could make the participant potentially non-compliant to the study procedures in the opinion of the Investigator.
* Mental condition rendering the participant or parent/guardian unable to understand the nature, scope, and possible consequences of the study.
* Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult or that would put the participant at risk by participating in the study in the opinion of the Investigator.
* History of drug or alcohol abuse.
* History of known human immunodeficiency virus (HIV) positivity.
* Pregnant or breast-feeding female participants or those who had planned to become pregnant during the study.
* Unwilling to agree to use a highly effective contraceptive method when receiving a course of alemtuzumab treatment and for 4 months following that course of treatment (fertile participants only).
* Female participants who have commenced menstruating (i.e., are of childbearing potential) and are unwilling or unable to be tested for pregnancy.
* Previous treatment with alemtuzumab.
* Treatment with natalizumab, daclizumab, fingolimod, methotrexate, azathioprine, cyclosporine, or mycophenolate mofetil in the last 6 months prior to screening, or determined by the treating physician to had residual immune suppression from these or other MS treatments.
* Treatment with teriflunomide in the last 12 months except if the participant underwent the recommended elimination procedure as per Summary of Product Characteristics (SmPC).
* Previous treatment with mitoxantrone, cyclophosphamide, cladribine, rituximab, ocrelizumab, leflunomide, or any cytotoxic therapy.
* Previous treatment with any investigational medication (drug that had not been approved at any dose or for any indication). Use of an investigational medication that is subsequently licensed and nonstandard use of a licensed medication (e.g., using a dose other than the dose that is stated in the licensed product labeling or using a licensed therapy for an alternative indication) was not exclusionary. Prior treatment with herbal medications or nutritional supplements was also permitted.
* Intolerance of pulsed corticosteroids, especially a history of steroid psychosis.
* History of malignancy.
* Prior documented history of thrombocytopenia, or platelet count at screening < lower limits of normal (LLN).
* Any disability acquired from trauma or another illness that, in the opinion of the Investigator, could interfere with evaluation of disability due to MS.
* Participants with known Type 1 hypersensitivity or anaphylactic reactions to the active substances or any of the excipients, or intolerance of acyclovir or its therapeutic equivalent.
* Major systemic disease or other illness that would, in the opinion of the Investigator, compromise participant safety or interfere with the interpretation of study results, e.g., current peptic ulcer disease, or other conditions that might predispose to hemorrhage, immune cytopenias, rheumatoid arthritis, systemic lupus erythematosus, other connective tissue disorders, vasculitis, inflammatory bowel disease, severe psoriasis.
* Medical, psychiatric, cognitive, or other conditions that, in the Investigator's opinion, compromise the participant's ability to understand the participant information, to give informed consent, to comply with the trial protocol, or to complete the study.
* Major psychiatric disorder that is not adequately controlled by treatment in the opinion of the Investigator.
* Epileptic seizures that are not adequately controlled by treatment.
* Magnetic resonance imaging (MRI)-related conditions: conditions that could interfere with MRI acquisition and/or interpretation of MRI results (eg, claustrophobia, orthopedic implants/treatments, orthodontic treatments etc).
* Known bleeding disorder (e.g., dysfibrinogenemia, factor IX deficiency, hemophilia, Von Willebrand's disease, disseminated intravascular coagulation, fibrinogen deficiency, clotting factor deficiency).
* Prior history of invasive fungal infections.
* Active infection, eg, deep-tissue infection, that the Investigator considers sufficiently serious to preclude study participation.
* In the Investigator's opinion, participant is at high risk for infection (e.g., indwelling catheter, dysphagia with aspiration, decubitus ulcer, history of prior aspiration pneumonia or recurrent urinary tract infection).

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2025-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (16):
- Investigational Site Number : 0400001, Vienna, Austria
- France (2):
  - Investigational Site Number : 2500001, Le Kremlin-Bicêtre
  - Investigational Site Number : 2500002, Strasbourg
- Italy (3):
  - Investigational Site Number : 3800004, Naples, Napoli
  - Investigational Site Number : 3800005, Cagliari
  - Investigational Site Number : 3800001, Milan
- Poland (3):
  - Investigational Site Number : 6160002, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160003, Lodz, Lódzkie
  - Investigational Site Number : 6160001, Warsaw
- Russia (4):
  - Investigational Site Number : 6430001, Moscow
  - Investigational Site Number : 6430004, Moscow
  - Investigational Site Number : 6430005, Saint Petersburg
  - Investigational Site Number : 6430002, Saint Petersburg
- Turkey (Türkiye) (2):
  - Investigational Site Number : 7920001, Ankara
  - Investigational Site Number : 7920003, Istanbul
- Investigational Site Number : 8260002, London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is being conducted at 21 sites in 10 countries. A total of 16 participants were screened and enrolled between 24-October-2017 and 07-September-2020.
Pre-assignment Details: Prior to alemtuzumab treatment phase (Month 0 to Month 8), participants underwent prior disease modifying therapy (DMT) phase during Month -4 to Month 0 (conducted to check participants eligibility for treatment). The DMT was discontinued 7 days prior to administration of first dose of alemtuzumab at Month 0. Data reported based on primary completion date of 04-May-2021.
Groups:
- Alemtuzumab: Participants with relapsing remitting multiple sclerosis (RRMS) underwent prior disease modifying therapy (DMT), from Month -4 to Month 0 (conducted to check participants eligibility for treatment) in prior DMT phase. After DMT phase, participants who were eligible for treatment, and with body weight greater than or equal to (>=) 50 kilograms (kg) received 12 milligrams per day (mg/day) of alemtuzumab, and participants with body weight less than (<) 50 kg received 0.24 milligrams per kilogram per day (mg/kg/day) of alemtuzumab administered as daily intravenous (IV) infusions at Month 0 for 5 consecutive days as first course of study treatment in alemtuzumab treatment phase.
Period: Phase1: Prior DMT:Month -4 to Month 0
Arm/Group | Alemtuzumab
Started | 16
Completed | 12
Not Completed | 4
Not completed — Physician Decision | 1
Not completed — Participant was withdrawn from study | 1
Not completed — Principal Investigator and Parents Decision | 1
Not completed — Still on Prior DMT Phase or missing Completion | 1
Period: Phase2:AlemtuzumabTreatment:Month 0 to 8
Arm/Group | Alemtuzumab
Started | 11 (Out of 12 participants who had completed Phase 1, one participant did not enter Phase 2.)
Treated | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on enrolled population.
Groups:
- Alemtuzumab: Participants with RRMS underwent prior DMT, from Month -4 to Month 0 (conducted to check participants eligibility for treatment) in prior DMT phase. After DMT phase, participants who were eligible for treatment, and with body weight >=50 kg received 12 mg/day of alemtuzumab, and participants with body weight <50 kg received 0.24 mg/kg/day of alemtuzumab administered as daily IV infusions at Month 0 for 5 consecutive days as first course of study treatment in alemtuzumab treatment phase.
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Brain Magnetic Resonance Imaging (MRI) Assessment: Number of New or Enlarged T2 Lesions Per MRI Scan
Description: Number of new or enlarged T2 lesions per scan was defined as the total number of new or enlarged T2 lesion that occurred during a specified period divided by the total number of scans performed during that specified period.
Time Frame: Period 1: Month -4 up to Month 0, Period 2: Month 4 to Month 8
Population: Analysis was performed on modified intent-to-treat (mITT) population that included participants who had received at least 1 dose of alemtuzumab and also had evaluable data for both Period 1 and Period 2. Data for this outcome measure was planned to be collected and analyzed separately for both periods.
Measure: Number (95% Confidence Interval); unit: lesions per scan
Groups:
- Period 1: Participants with RRMS who were assessed from Month -4 up to Month 0 (prior DMT phase) to confirm their eligibility for the administration of alemtuzumab IV infusion at Month 0. A baseline magnetic resonance imaging (MRI) was performed close to Month -4 during the screening period and another at Visit 3 (in between Day -14 to Day -7). Both MRI were taken while participants were on their prior DMT. It was important to ensure that these 2 MRI assessments were performed 4 months (±7 days) apart.
- Period 2: Participants with RRMS and with body weight >=50 kg received 12 mg/day of alemtuzumab, and participants with body weight <50 kg received 0.24 mg/kg/day alemtuzumab administered as daily IV infusions at Month 0 for 5 consecutive days as first course of study treatment. Period 2 occurred from Month 4 to Month 8. The MRI performed at the Month 4 visit was the baseline MRI for Period 2. A second MRI was performed after alemtuzumab first course of treatment at Month 8. It was important to ensure that these 2 MRI assessments were performed 4 months (±7 days) apart.
Arm/Group | Period 1 | Period 2
Number analyzed (Participants) | 11 | 11
lesions per scan | 3.53 [1.78 to 7.03] | 0.13 [0.03 to 0.48]

2. Secondary Outcome: Brain Magnetic Resonance Imaging (MRI) Assessment: Number of Participants With New or Enlarged T2 Lesions Per MRI Scan
Description: Number of participants with at least one new or enlarged T2 lesions per MRI scan was reported in this outcome measure. Number of new or enlarged T2 lesions per scan was defined as the total number of new or enlarged T2 lesion that occurred during treatment period divided by the total number of scans performed during treatment period.
Time Frame: Period 1: Month -4 up to Month 0, Period 2: Month 4 to Month 8
Population: Analysis was performed on mITT population. Data for this outcome measure was planned to be collected and analyzed separately for both periods.
Measure: Count of Participants; unit: Participants
Groups:
- Period 1: Participants with RRMS who were assessed from Month -4 up to Month 0 (prior DMT phase) to confirm their eligibility for the administration of alemtuzumab IV infusion at Month 0. A baseline MRI was performed close to Month -4 during the screening period and another at Visit 3 (in between Day -14 to Day -7). Both MRI were taken while participants were on their prior DMT. It was important to ensure that these 2 MRI assessments were performed 4 months (±7 days) apart.
Arm/Group | Period 1 | Period 2
Number analyzed (Participants) | 11 | 11
Participants | 10 | 3

3. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Score at Months 4 and 8
Description: EDSS is an ordinal scale in half-point increments that qualifies disability in participants with MS. It consists of 8 ordinal rating scales assessing seven functional systems (pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral, and other). EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS), where higher scores indicated worst outcomes.
Time Frame: Baseline, Months 4 and 8
Population: Analysis was performed on mITT population. Here, 'number analyzed' signifies participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 11
scores on scale
  Month 4 | 0.05 (0.52)
  Month 8 | 0.00 (0.55)

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE) and Treatment-emergent Serious Adverse Events (TESAE)
Description: Data for this outcome measure will be reported at the time of anticipated last participant last visit results posting (December 2026).
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-12

5. Secondary Outcome: Annualized Relapse Rate (ARR)
Description: as for outcome 4
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-12

6. Secondary Outcome: Change From Baseline in Cognition Test Scores of Brief Visuospatial Memory Test - Revised (BVMT-R)
Description: as for outcome 4
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-12

7. Secondary Outcome: Change From Baseline in Cognition Test Scores of Symbol Digit Modality Test (SDMT)
Description: as for outcome 4
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-12

8. Secondary Outcome: Change From Baseline in Quality of Life (QoL) Measures of Pediatric Quality of Life (PedsQL) Questionnaire Score
Description: as for outcome 4
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-12

9. Secondary Outcome: Change From Baseline in Pediatric Quality of Life in Neurological Disorders (NeuroQoL) Questionnaire Score
Description: as for outcome 4
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-12

10. Secondary Outcome: Serum Concentrations of Alemtuzumab Over Time
Description: as for outcome 4
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-12

11. Secondary Outcome: Maximum Serum Concentration Observed (Cmax) of Alemtuzumab
Description: as for outcome 4
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-12

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Alemtuzumab
Description: as for outcome 4
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-12

13. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) of Alemtuzumab
Description: as for outcome 4
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-12

14. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-last) of Alemtuzumab
Description: as for outcome 4
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-12

15. Secondary Outcome: Terminal Half-life (T1/2z) of Alemtuzumab
Description: as for outcome 4
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-12

16. Secondary Outcome: Assessment of Lymphocyte Phenotyping
Description: as for outcome 4
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-12

17. Secondary Outcome: Percentage of Participants With Incidence of Antidrug Antibodies (ADA)
Description: as for outcome 4
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: All reported AEs were collected from Month -4 up to Month 0 for prior DMT Phase; and from first dose of alemtuzumab (Month 0) up to 8 months for alemtuzumab treatment phase
Groups:
- Prior DMT Phase: Participants with RRMS were assessed from Month -4 up to Month 0 in prior DMT phase to confirm their eligibility for the administration of alemtuzumab IV infusions in alemtuzumab treatment phase.
- Alemtuzumab: After DMT phase, participants who were eligible for treatment, and with body weight >=50 kg received 12 mg/day of alemtuzumab, and participants with body weight <50 kg received 0.24 mg/kg/day of alemtuzumab administered as daily IV infusions at Month 0 for 5 consecutive days as first course of study treatment in alemtuzumab treatment phase.
Arm/Group | Prior DMT Phase | Alemtuzumab
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/11
Serious Adverse Events (participants affected / at risk) | 3/16 | 3/11
Other Adverse Events (participants affected / at risk) | 10/16 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prior DMT Phase (N=16) | Alemtuzumab (N=11)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 1 (1)
Multiple Sclerosis Relapse (Nervous system disorders) | 3 (4) | 1 (1)
Uhthoff's Phenomenon (Nervous system disorders) | 1 (1) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prior DMT Phase (N=16) | Alemtuzumab (N=11)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 3 (4)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (6)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces Discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Paraesthesia Oral (Gastrointestinal disorders) | 0 (0) | 1 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest Discomfort (General disorders) | 0 (0) | 1 (3)
Discomfort (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 5 (7)
Influenza Like Illness (General disorders) | 1 (1) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 2 (3)
Oedema Peripheral (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Peripheral Swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 5 (10)
Mite Allergy (Immune system disorders) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Genitourinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (4) | 6 (7)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection Viral (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 3 (3) | 3 (5)
Tinea Versicolour (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 3 (6)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Viral Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Blood Urine (Investigations) | 0 (0) | 1 (1)
Heart Rate Increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 0 (0) | 1 (1)
Weight Increased (Investigations) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendon Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (3)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 6 (17)
Multiple Sclerosis Relapse (Nervous system disorders) | 3 (4) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (3)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sensory Disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Uhthoff's Phenomenon (Nervous system disorders) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Fear (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Sleep Disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT03368664/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT03368664/SAP_001.pdf